CLINICAL TRIAL: NCT06515548
Title: Assessment the Efficacy of Vitamin D Mouth Rinse Versus Placebo in the Treatment of Molar Incisor Hypomineralization In Vitro Study and in Situ Randomized Double-Blind Placebo Controlled Clinical Trial.
Brief Title: Assessment the Efficacy of Vitamin D Mouth Rinse Versus Placebo in the Treatment of MIH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: MTI University (Other)
Responsible Party: Principal Investigator, Parryhan Mohamed Abdelsamie, Lecturer of periodontology, MTI University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PMTIU
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Molar Incisor Hypomineralization
Keywords: vitamin D; MIH; vitamin D mouth rinse; Molar Incisor Hypomineralization; vitamin D mouthwash; Topical vitamin D
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Intervention Model Description: In vitro study and in situ Randomized Double-Blind Placebo controlled Clinical Trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: Double-Blind Placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D mouthwash (Active Comparator): a
  Interventions: Drug: Vitamin D3 mouth wash
- Placebo mouth wash (Placebo Comparator)
  Interventions: Drug: Vitamin D3 mouth wash

INTERVENTIONS:
Drug: Vitamin D3 mouth wash — topical vitamin D oral mouth wash as every 10ml of the solution contains 3000 IU
  Other Names: Vitamin D3 mouth rinse

SUMMARY:
In child patients with molar incisor hypo mineralization, Will Vitamin D mouth wash offer more success for patients with MIH as regards better MIH TNI index, decrease plaque accumulation, more gingival health and less bleeding on probing differentiated from placebo mouthwash?

DETAILED DESCRIPTION:
Molar incisor hypomineralization (MIH) refers to specific developmental qualitative defect of the enamel that typically affect 1 to all 4 of the permanent molars and can also involve the permanent incisors.

MIH is clinically characterized by morphological enamel defects that can be seen on the occlusal surface of permanent molars and the incisal one-third (or more) of the incisors result from hypomineralization. These defects more or less well-defined opacities that vary in size and can be discoloured from white to yellow brownish. The hypomineralized enamel is friable and has inferior mechanical properties as well as reduced modulus of elasticity when compared to sound enamel.

As a consequence, hypomineralized enamel leads to post-eruptive breakdown and hypersensitivity, and it is prone to development of carious lesions and pain. Due to pain, fragile enamel and increased treatment need at an early point of time in life, MIH treatment represents a clinical challenge. The well-defined opacities are focal subsurface decalcifications in enamel are commonly associated with extended plaque retention. Periodontal disease in children is mainly limited to gingival inflammation and is observed as gingival oedema, colour and contour changes, bleeding on probe or spontaneous bleeding.

Recent study showed that plaque accumulation and gingival inflammation were higher in patients with MIH compared with healthy children, and that oral hygiene and gingival health worsened as the severity of MIH increased.

Vitamin D, plays a pivotal role in many biological functions such as in innate immunity effect, the regulation of calcium (Ca+) and phosphate metabolism and their deposition in mineralized tissues. Since the presence of Vitamin D3 receptors on ameloblast and odontoblast cells, its function in tooth development and remineralization, changes in the biochemical composition of saliva and immunological modulation of dental infection has been suggested.

Vitamin D has been demonstrated to have significant potential in improving the remineralization of early lesions on enamel surfaces enhancing surface microhardness and minerals content. Remineralization is defined as the process whereby calcium and phosphate ions are supplied from a source external to the tooth to promote ion deposiption into crystal voids in demineralized enamel, to produce net mineral gain.

Recent ex-vivo study revealed that the topical application of fluoride and vitamin D promoted the formation of persistent mineral crystals on enamel surfaces of deciduous teeth. Consequently, this study recommends further evaluation to be potentially used as an alternative strategy.

The treatment of teeth affected by MIH should be a minimally invasive procedure that aims to protect, strengthen and preserve dental structure. Numerous therapeutic alternatives have been proposed over time for the treatment of MIH-affected teeth, but the clinical management of these conditions is very demanding and less conservative.

ELIGIBILITY:
Inclusion Criteria:

1. More than 6 years' child with all permanent incisors and first molar teeth are fully erupted with all surfaces visible.
2. At least one affected first permanent molar were considered to have MIH (Lygidakis et al. 2010; Kühnisch et al. 2014).
3. No chronic systemic disease
4. No acute infection
5. cooperative Child

Exclusion Criteria:

1. Drugs (chlorhexidine-based gels and mouthwashes)
2. Hypomineralization with a diameter less than 1 mm.
3. Hypoplastic defects, fluorosis (diffuse hypomineralization), amelogenesis imperfecta, and dentinogenesis imperfecta.
4. Defects on approximal surfaces and diffuse opacities.
5. Fixed orthodontic treatment

   -

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2024-08-30 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
MIH TNI | 3 months
Gingival Index | 3 months
Plaque Index | 3 months

SECONDARY OUTCOMES:
Bleeding on Probing | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Parryhan M Abdelsamie, PhD, Principal Investigator — MTI University
Locations (1):
- Cairo University, Faculty of Dentistry., Giza, Egypt

IPD SHARING:
Plan to Share IPD: No